CLINICAL TRIAL: NCT06696482
Title: Effort and Antidepressant Study Test
Acronym: EAST
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EAST_Study
Record Dates: First submitted 2024-11-15; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Effort Based Decision Making; Prosocial Behavior; Apathy
Keywords: fMRI
MeSH Terms: conditions — Altruism; Lethargy | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Escitalopram (Experimental): Escitalopram tablets 10 mg once daily for 7 days
  Interventions: Drug: Escitalopram 10mg
- Placebo (Placebo Comparator): Lactose tablets 10 mg once daily for 7 days
  Interventions: Drug: Placebo 10 mg

INTERVENTIONS:
Drug: Escitalopram 10mg — Escitalopram 10 mg, encapsulated in an opaque capsule to facilitate blinding of participant and researcher
  Arms: Escitalopram
Drug: Placebo 10 mg — Placebo 10 mg, encapsulated in an opaque capsule to facilitate blinding of participant and researcher
  Arms: Placebo

SUMMARY:
The aim of this study is to investigate the behavioural effects and neural correlates of increasing serotonin levels in healthy volunteers, through a 7-day course of the SSRI escitalopram, on an effort-based decision-making task measuring self-benefiting and prosocial behaviours.

DETAILED DESCRIPTION:
This study investigates the mechanisms behind motivation and apathy, focusing on how effort is dedicated to both self-benefiting and prosocial actions. Diminished motivation, often manifesting as apathy, is associated with poor health outcomes and is common in neurological disorders like Parkinson's, Alzheimer's, and small vessel cerebrovascular disease (SVD). While brain regions like the dorsal anterior cingulate cortex (dACC), dorsomedial prefrontal cortex (dmPFC), and anterior insula (AI) are known to regulate motivation in reward-based decision-making for personal gain, prosocial motivation remains underexplored. Prosocial behaviour involves actions that benefit others and contribute to physical and psychological well-being. Recent studies suggest unique neural activity in the anterior cingulate gyrus (ACCg) during prosocial actions, differing from self-benefiting behaviour.

To the best of our knowledge, there is no prior evidence on how SSRIs might influence prosocial motivation or its neural correlates. This study will address this gap by examining SSRI effects on effort-based prosocial decision-making, potentially identifying novel insights into the neural mechanisms underlying motivation for prosocial behaviour.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the research
* Aged 18 to 40 years
* Sufficient knowledge of English language to understand and complete study tasks
* Right-handed

Exclusion Criteria:

* Current or past probable diagnosis of psychiatric illness, according to DSM-5 criteria requiring intervention by a healthcare professional, including but not limited to psychosis, bipolar disorder, major depression, OCD, PTSD, substance abuse disorder or any eating disorder
* Current or past diagnosis of any significant personality disorder (e.g., borderline personality disorder) according to self-report
* Diagnosis of attention deficit hyperactive disorder or autistic spectrum disorder that impairs daily functioning, requires pharmacotherapy or in the opinion of the study medic would affect the scientific integrity of the study
* Current use of medication that might interact with the effects of escitalopram or affect the scientific integrity of the study
* Previous suicide attempt or previous prolonged period (eg., > 5 days) of thought to end life
* Known contraindication to escitalopram including: past allergic reaction to escitalopram or any other medicines, diagnosis of angle-closure glaucoma, or current use of any other medication whose use interacts with escitalopram (according to BNF guidance) e.g. associated with prolonged QT-interval
* Any other current or past medical conditions which in the opinion of the study medic may interfere with the safety of the participant or the scientific integrity of the study including epilepsy/seizures, brain injury, hepatic or renal disease, diabetes, severe gastro-intestinal problems, Central Nervous System (CNS) tumours, neurobiological conditions
* First-degree relative with a diagnosis of schizophrenia-spectrum or other psychotic disorder, or bipolar disorder
* Severely underweight (BMI<17) or very obese (BMI>40) in a manner that renders them unsuitable for the study in the opinion of the study medic
* Heavy use of cigarettes (smoke>20 cigarettes per day)
* Heavy use of caffeine (drink>4 x 250 ml cups/cans of coffee/energy drinks per day)
* Lactose intolerance (due to the study involving administration of a lactose placebo tablet)
* Pregnancy (as determined by urine pregnancy test taken during the Part 2 screening visit), breast feeding or plans to become pregnant
* Past history of dependence on illicit substances or regular illicit substances use within the previous three months
* Evidence of current or past harmful use of alcohol
* Previous participation in a study involving the tasks used in this study or involving use of escitalopram in the last year in the Department of Psychiatry (University of Oxford)
* Physical (including visual and auditory) or language impairment that would make complying with the study protocol challenging.
* Participant is unlikely to comply with the clinical study protocol or is unsuitable for any other reason, in the opinion of the investigator
* Not suitable for MRI neuroimaging, e.g., difficulty remaining still for duration of scan
* Any MRI contraindications outlined in FMRIB 3 Tesla scanning safety form

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Effort-based decision-making task for self-benefiting and prosocial behaviours: behavioural correlates | Day 7 of treatment
  In the fMRI scanner task, participants are prompted to choose between two offers on each trial. One option allows them to earn a low reward for minimal effort (rest), while the other presents a variable higher-reward, higher-effort (work) of the same duration. The low-reward, low-effort offer earns 1 point without exertion. Higher-reward, higher-effort offers range from 2 to 10 points (in 2-point-increments) and effort varies from 30% to 70% (in 10% increments) of their MVC.
  Each trial differs in whether the outcome is delivered to the participant themselves (self) or someone else (prosocial). Effort levels for each offer are visually represented using coloured portions of a pie chart and rewards (points) are displayed in colour below.
Effort-based decision-making for self-benefiting and prosocial behaviours: Neural correlates | Day 7 of treatment
  Activity of brain regions associated with self-benefiting and prosocial behaviours

SECONDARY OUTCOMES:
Emotional processing: Faces task | Day 7 of treatment
  During the emotional processing face task participants will be presented with pictures of emotional faces and asked to label the emotions into different categories.
Prosocial behaviour: Social learning task | Day 7 of treatment
  This game involves making fictitious investment decisions with other "previous participants in our lab" (programmed responses) and trying to maximize the number of points earned in the game.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine J Harmer, PhD, Principal Investigator — University of Oxford

IPD SHARING:
Plan to Share IPD: Undecided
Research data will be anonymised and then processed for analysis. Anonymised data will be made available post-publication on Open Science Framework (OSF).
  we plan to share normalised MRI data (such that unique brain structure is not shared) into an online scientific data sharing repository such as 'Zenodo'